CLINICAL TRIAL: NCT03202628
Title: Phase 2 Trial of Induction With Ixazomib, Pomalidomide, Dexamethasone Prior to Salvage Autologous Stem Cell Transplant Followed by Consolidation With Ixazomib, Pomalidomide, and Dexamethasone and Ixazomib Maintenance in Multiple Myeloma
Brief Title: Ixazomib Citrate, Pomalidomide, Dexamethasone, Stem Cell Transplant in Treating Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC168A; NCI-2017-01145 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC168A (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; ixazomib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib, pomalidomide, dexamethasone, ASCT) (Experimental): INDUCTION (COURSES 1-4): Patients receive ixazomib citrate PO on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days (courses 1-3) and 56 days (course 4) for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  TRANSPLANTATION (COURSE 5): Between 2-4 weeks following Induction, patients undergo ASCT.
  CONSOLIDATION (COURSES 6-9): Beginning 60-120 days following ASCT, patients receive ixazomib citrate, pomalidomide, and dexamethasone as in Induction. Treatment repeats every 28 days (courses 6-8) and 56 days (course 9) for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE (COURSES 10+): Beginning 0-4 weeks following Consolidation, patients receive ixazomib citrate as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Dexamethasone; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Drug: Pomalidomide

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: autologous stem cell transplantation
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II trial studies how well ixazomib citrate, pomalidomide, dexamethasone, and stem cell transplantation works in treating patients with multiple myeloma that has come back or does not respond to treatment. Giving chemotherapy, such as pomalidomide and dexamethasone, before a stem cell transplant helps kill any cancer cells that are in the body and helps make room in the patient?s bone marrow for new blood-forming cells (stem cells) to grow. After treatment, stem cells are collected from the patient's blood and stored. More chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving ixazomib citrate in addition to pomalidomide, dexamethasone, and stem cell transplantation may work better in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of progression free survival at 18 months from study entry after therapy with ixazomib citrate (ixazomib [MLN9708]) in combination with pomalidomide and dexamethasone followed by a single autologous stem cell transplantation (ASCT) and consolidation with ixazomib in combination with pomalidomide and dexamethasone and maintenance with ixazomib in relapsed refractory ASCT naive multiple myeloma (MM) patients.

SECONDARY OBJECTIVES:

I. To determine the best overall response rates (>= partial response [PR]) and deep responses (very good partial response [VGPR], complete response [CR], stringent complete response [sCR]) at various stages of treatment: after induction, after stem cell transplantation (SCT), after consolidation and during maintenance.

II. To determine the overall survival from study entry.

TERTIARY OBJECTIVES:

I. Assessment of minimal residual disease (MRD) by flow cytometry at various stages of treatment: after induction, day # 100 after SCT, after consolidation and during maintenance at year 1 and 2 from initiation of maintenance therapy.

II. To determine the engraftment kinetics (white blood cells [WBC] and platelet) following single salvage ASCT for relapsed disease.

OUTLINE:

INDUCTION (COURSES 1-4): Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15, pomalidomide (PO) on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days (courses 1-3) and 56 days (course 4) for up to 4 courses in the absence of disease progression or unacceptable toxicity.

TRANSPLANTATION (COURSE 5): Between 2-4 weeks following Induction, patients undergo ASCT.

CONSOLIDATION (COURSES 6-9): Beginning 60-120 days following ASCT, patients receive ixazomib citrate, pomalidomide, and dexamethasone as in Induction. Treatment repeats every 28 days (courses 6-8) and 56 days (course 9) for up to 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE (COURSES 10+): Beginning 0-4 weeks following Consolidation, patients receive ixazomib citrate as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until progressive disease, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated ASCT naive MM patients, currently with relapsed or refractory disease who are being considered for single ASCT for relapsed disease; patients must be eligible to undergo a stem cell transplant as per institutional criteria for selection at the time of registration
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 75 x 10^9/L unless the participant has >= 50% bone marrow infiltration in which case a platelet count of >= 50 x 10^9/L is allowed
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x the upper limit of the normal range (ULN) or if total bilirubin is > 1.5 x ULN, the direct bilirubin must be =< 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN or < 5 x ULN if liver involvement
* Patients with measurable disease defined as at least one of the following:

  * Serum monoclonal protein >= 1.0 g/dL by protein electrophoresis
  * >= 200 mg of monoclonal protein in the urine on 24-hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Willing to provide informed written consent
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Willing to follow strict birth control measures
* Persons of childbearing potential, agree to one of the following:

  * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Persons able to father a child: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to follow the requirements of the Pomalyst REMS program
* Willing to return to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide bone marrow samples under Institutional Review Board (IRB)#521-93 for correlative research purposes

Exclusion Criteria:

* Diagnosed or treated for another malignancy =< 2 years prior to registration or previously diagnosed with another malignancy and have any evidence of residual disease

  * NOTE: If there is a history or prior malignancy, patient must not be receiving other specific treatment for their cancer; patients with non-melanoma skin cancer or carcinoma in situ of any type, or low-risk prostate cancer after curative therapy, are not excluded if they have undergone complete resection
  * NOTE: Platelet transfusions to help patients meet eligibility criteria are not allowed =< 3 days prior to study registration
* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens; NOTE: this includes uncompensated heart or lung disease
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm; NOTE: Bisphosphonates are considered to be supportive care rather than therapy and are allowed while on protocol treatment
* Patient has >= grade 2 peripheral neuropathy, or grade 1 with pain on clinical examination during the screening period
* Major surgery =<14 days prior to registration
* Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or use of Ginkgo biloba or St. John?s wort =< 14 days prior to registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. NOTE: Any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Corrected QT (QTc) > 470 milliseconds (msec) on a 12-lead ECG obtained during the screening period; Note: If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG
* Known human immunodeficiency virus (HIV) positive
* Known hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Known allergy to any of the study medications, their analogues or excipients in the various formulations
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of study treatment including difficulty swallowing
* Diarrhea > grade 1, based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0 grading, in the absence of antidiarrheals
* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior chemotherapy
* Radiotherapy =< 14 days prior to registration; NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Central nervous system involvement with disease under study (myeloma), or concurrent AL amyloidosis or plasma cell leukemia
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not
* Prior stem cell transplantation for myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Kapoor, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT): INDUCTION (COURSES 1-4): Patients receive ixazomib citrate PO on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days (courses 1-3) and 56 days (course 4) for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  >
  > TRANSPLANTATION (COURSE 5): Between 2-4 weeks following Induction, patients undergo ASCT.
  >
  > CONSOLIDATION (COURSES 6-9): Beginning 60-120 days following ASCT, patients receive ixazomib citrate, pomalidomide, and dexamethasone as in Induction. Treatment repeats every 28 days (courses 6-8) and 56 days (course 9) for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  >
  > MAINTENANCE (COURSES 10+): Beginning 0-4 weeks following Consolidation, patients receive ixazomib citrate as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Autologous Hematopoietic Stem Cell Transplantation: Undergo ASCT
  >
  > Dexamethasone: Given PO
  >
  > Ixazomib Citrate: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Pomalidomide: Given PO
Period: Overall Study
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT): INDUCTION (COURSES 1-4): Patients receive ixazomib citrate PO on days 1, 8, and 15, pomalidomide PO on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days (courses 1-3) and 56 days (course 4) for up to 4 courses in the absence of disease progression or unacceptable toxicity.> > TRANSPLANTATION (COURSE 5): Between 2-4 weeks following Induction, patients undergo ASCT.>
  > CONSOLIDATION (COURSES 6-9): Beginning 60-120 days following ASCT, patients receive ixazomib citrate, pomalidomide, and dexamethasone as in Induction. Treatment repeats every 28 days (courses 6-8) and 56 days (course 9) for up to 4 courses in the absence of disease progression or unacceptable toxicity.>
  > MAINTENANCE (COURSES 10+): Beginning 0-4 weeks following Consolidation, patients receive ixazomib citrate as in Induction. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Autologous Hematopoietic Stem Cell Transplantation: Undergo ASCT>
  > Dexamethasone: Given PO>
  > Ixazomib Citrate: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Pomalidomide: Given PO
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Revised international staging system (R-ISS) myeloma stage at initial diagnosis [Count of Participants; unit: Participants] — Stage I (All criteria must be met) - Serum β2 microglobulin<3.5 mg/L; Serum albumin≥3.5 g/dL; Del(17p) and/or t(4;14) and/or t(14;16)=No; Abnormal LDH level=No
  Stage II - All other possible combinations (not Stage I or Stage III)
  Stage III (All criteria must be met) - Serum β2 microglobulin>5.5 mg/L; Serum albumin=NA; Del(17p) and/or t(4;14) and/or t(14;16)=Yes AND/OR Abnormal LDH level=Yes
  The higher the stage, the worse the prognosis.
  Participants
    Stage I | 2
    Stage II | 5
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 18 Months (PFS18) Defined as the Proportion of Patients Alive and Free From Disease Progression at 18 Months From Study Entry
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success proportion will be calculated. If patients are censored prior to 18 months post registration, a Kaplan Meier (Kaplan, E. and Meier, P., 1958) estimate for PFS18 along with the 95% confidence intervals will be reported.
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
proportion of participants | 0.3750 [0.0852 to 0.7551]

2. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) Very Good Partial Response (VGPR) Rate
Description: Will be estimated by the number of patients who achieve a stringent complete response (sCR), complete response CR, or VGPR divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall >= VGPR will be calculated.
Time Frame: 30 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
percentage of patients | 25 [3.19 to 65.09]

3. Secondary Outcome: Number of Patients Experiencing Adverse Events Graded According to the Medical Dictionary for Regulatory Activities (MedDRA) Version (v) 12.1
Description: The number of patients experiencing a grade 3 or greater adverse event will be reported. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
Participants | 7

4. Secondary Outcome: Overall Response Rate
Description: Will be estimated by the number of patients who achieve a stringent complete response (sCR), complete response CR, very good partial response (VGPR), or partial response (PR) divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true overall response rate will be calculated.
Time Frame: 30 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
percentage of patients | 50 [15.7 to 84.3]

5. Secondary Outcome: Percent of Patients Alive at 30 Months
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: 30 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
Number analyzed (Participants) | 8
percentage of patients | 75 [50.3 to 100]

6. Other Pre Specified Outcome: Change in Minimal Residual Disease (MRD) in Bone Marrow Assessed by Flow Cytometry
Description: The proportion of patients who achieve MRD negative status will be estimated by the number of patients who are MRD negative divided by the total number of evaluable patients who achieve a stringent complete response (sCR) or complete response (CR). Exact binomial 95% confidence intervals for the true MRD negative rate will be calculated.
Time Frame: Baseline up to 1 year from initiation of maintenance therapy
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Engraftment Kinetics (White Blood Cells [WBC] and Platelet) Following Single Salvage Autologous Stem Cell Transplantation (ASCT)
Description: Will be measured by assessing the timing of recovery of bone marrow function. Will be summarized using descriptive statistics.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT)
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT) (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib, Pomalidomide, Dexamethasone, ASCT) (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (33)
Diarrhea (Gastrointestinal disorders) | 6 (61)
Nausea (Gastrointestinal disorders) | 4 (25)
Vomiting (Gastrointestinal disorders) | 1 (3)
Fatigue (General disorders) | 8 (50)
Urinary tract infection (Infections and infestations) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 4 (13)
Lymphocyte count decreased (Investigations) | 6 (30)
Neutrophil count decreased (Investigations) | 8 (23)
Platelet count decreased (Investigations) | 7 (16)
White blood cell decreased (Investigations) | 8 (26)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (61)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT03202628/Prot_SAP_000.pdf